CLINICAL TRIAL: NCT05540639
Title: Development and Evaluation of Somali-adapted Mindfetalness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sophiahemmet University (Other)
Collaborators: Karolinska Institutet (Other); Dalarna University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: Somali-adapted Mindfetalness
Record Dates: First submitted 2022-06-30; First posted 2022-09-15 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2024-11

CONDITIONS: Prevention

STUDY DESIGN:
Intervention Model Description: Pregnant women born in Somalia with singleton pregnancy
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention with modified Mindfetalness (Experimental): The pregnant woman will be informed about the possibility of practicing Mindfetalness verbally, by a video, in a leaflet and at a website. The practice is described as spending 15 minutes every day from gestational week 28+0 to get to know the fetal movement pattern. The fetus must be awake when practicing Mindfetalness and the woman is suggested to lay on her left side when she observes fetal movements. In the leaflet the woman can write down something about the nature, frequency or strength of the fetal movements. If the woman experiences decreased frequency of fetal movements or weaker movements she is instructed to seek healthcare without unnecessary delay.
  Interventions: Behavioral: Modified Mindfetalness
- Routine care (No Intervention): Historical comparison of the maternal clinics before the intervention. No activities have been taken place.

INTERVENTIONS:
Behavioral: Modified Mindfetalness — The pregnant woman is motivated to practice Mindfetalness verbally, by video, by a leaflet and at a website.
  Arms: Intervention with modified Mindfetalness

SUMMARY:
Development of Somali-adapted Mindfetalness: Interviews with women born in Somalia

A before-after study:

Intervention: pregnant women receive a pamphlet, introduction to Mindfetalness by her midwife during the gestational-week 25 visit. The pregnant woman will well get access to a website concerning Mindfetalness. The pregnant women will be encouraged to start practicing Somali-adapted Mindfetalness during gestational week 28.

Comparison: Intervention period (1/1-2022 to 31/12 2023) compared to 5 years before (1/1 2015 to 31/12 2019)

DETAILED DESCRIPTION:
Development of Somali-adapted Mindfetalness, initial data collection:

Pregnant women or recently given birth. Women born in Somalia with a singleton pregnancy from gestational week 28+0. Interviews focusing on fetal movements, reactions to fetal movements, and facilitating and inhibiting factors for seeking care for pregnancy-related conditions will be carried out. After transcription verbatim, the text will be analyzed with modified content analysis as described by Elo & Kyngäs.

A before-after study:

Population: Women born in Somalia registered at one of the 31 antenatal clinics where under 2019 ten or more women were registered. The registration will be either 1/1 2022 to 31/12 2023 or 1/1 2015 and 31/12 2019 (1/1 2020 to 31/12 2021 has been omitted to diminish a possible confounding effect of the COVID-19 pandemic.)

Intervention: In the chosen 31 antenatal clinics, midwives will receive an education in Somali-adapted Mindfetalness. Moreover, each pregnant woman registered after 1/1 2022 and before 31/12 2023, will receive a pamphlet, introduction to Mindfetalness by her midwife during the gestational-week 25 visit. The pregnant woman will well get access to a website concerning Mindfetalness. The pregnant women will be encouraged to start practicing Somali-adapted Mindfetalness during gestational week 28.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman living in Sweden but born in Somalia, in gestational age minimum 24+0

Exclusion Criteria:

* None

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 5628 (Actual)
Dates: Start 2022-01-11 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Seeking care due to decreased fetal movements | From pregnancy week 22+0 until birth
  The investigators will use the ICD-code (International Classification of Diseases) AM041 (examination due to decreased fetal movements) where applicable
  . The Investigators will use the data from The Swedish Pregnancy Register.
Apgar score <10 | At delivery, five minutes after birth
  The investigators will use the information reported to the Swedish Pregnancy Register.
Apgar score <7 | At delivery, five minutes after birth
  The investigators will use the information reported to the Swedish Pregnancy Register.

SECONDARY OUTCOMES:
Induction of labour | At delivery
  The investigators will use the information reported to the Swedish Pregnancy Register. The responsible healthcare professionals classify mode of delivery and report it to the register. The register is population-based and covers by and large every birth in the region at the time.
Cesarean section (planned) | At delivery
  The investigators will use the information reported to the Swedish Pregnancy Register. The responsible healthcare professionals classify mode of delivery and report it to the register. The register is population-based and covers by and large every birth in the region at the time.
Cesarean section (emergency) | At delivery
  The investigators will use the information reported to the Swedish Pregnancy Register. The responsible healthcare professionals classify mode of delivery and report it to the register. The register is population-based and covers by and large every birth in the region at the time.
Transfer to Neonatal Intensive Care Unit (NICU) | At delivery
  The investigators will use the Swedish Neonatal Quality Register. The responsible healthcare professionals report transfer to NICU to the register. The register is population-based and covers by and large every birth in the region at the time.

OTHER OUTCOMES:
Apgar score <4 | At delivery, five minutes after birth
  The investigators will use the information reported to the Swedish Pregnancy Register.
Spontaneous start of labour | At delivery
  The investigators will use the information reported to the Swedish Pregnancy Register. The responsible healthcare professionals classify mode of delivery and report it to the register. The register is population-based and covers by and large every birth in the region at the time.

CONTACTS AND LOCATIONS:
Locations (1):
- Ingela Rådestad, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-02-11): https://cdn.clinicaltrials.gov/large-docs/39/NCT05540639/SAP_001.pdf